CLINICAL TRIAL: NCT02686944
Title: A Phase I Open-label Study Evaluating Safety and Efficacy of Intratumorally Administered Intuvax in Patients With Progressing Gastrointestinal Stromal Tumors (GIST) During Ongoing Second, Third or Fourth Line Treatment With Tyrosine Kinase Inhibition Therapy. A Prospective Single Armed, Open Label Phase I Safety and Efficacy Study
Brief Title: A Study to Evaluate the Safety of Intuvax Administered Intra-tumorally in Patients With Gastrointestinal Stromal Tumors
Acronym: GIST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mendus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-103; 2015-002689-22 (EudraCT Number)
Record Dates: First submitted 2016-01-19; First posted 2016-02-22 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Intuvax (ilixadencel) (Experimental): Intuvax (ilixadencel) will be administered 2 or 3 times. First injection Day 1 (pat 1-12), second injection 14 days after the first vaccination (pat 1-12), third injection 28 days after the second vaccination (only pat 7-12).
  Max 10 000 000 allogeneic dendritic cells/ml per injection.
  Interventions: Biological: Intuvax (ilixadencel)

INTERVENTIONS:
Biological: Intuvax (ilixadencel) — Therapeutic vaccine: allogeneic, proinflammatory dendritic cells, suspension for intratumoral injection
  Other Names: ilixadencel

SUMMARY:
The study is a prospective single armed, open label phase I study. Patients with advanced or metastatic GIST and tumor progression despite ongoing treatment with second, third or fourth line TKI treatment, and with at least one measureable tumor lesion, will be eligible for the study. A maximum of 12 patients will be included in this study. The patients will continue with TKI treatment until the 3 months follow up visit. If further tumor progression TKI will be withdrawn but if stable disease or objective response the patient will continue with TKI until progress. The investigational product Intuvax will be injected into a tumor lesion at two or three treatment occasions; day 1, 14 days (±3 days) after the first vaccination, and 28 days (±3 days) after the second vaccination (patient 7-12 only). Intuvax will be injected in a viable part of the tumor, using ultrasound-guided or CT technique for correct administration.

ELIGIBILITY:
Inclusion Criteria:

1. Be informed of the nature of the study and have provided written informed consent.
2. At least 18 years of age.
3. Diagnosis of GIST (according to modified NIH criteria, 2011) where curative excision is no longer an option, i.e. confirmed unresectable or metastatic GIST, and that has progressed on second, third or fourth line tyrosine kinase inhibitor (TKI) treatment.
4. Radiologically measurable tumor(s), i.e at least 3 cm in longest uni-dimensional diameter as measured by CT
5. Clinical and/or CT verified disease progression despite ongoing second, third or fourth line treatment with a TKI
6. Female who has been post-menopausal for more than one (1) year or female of childbearing potential using a highly efficient method of contraception (i.e. a method with less than 1% failure rate [e.g. sterilization, hormone implants, hormone injections, some intrauterine devices, or vasectomized partner with combined use of condom and/or birth control pills]) during study participation. Female of childbearing potential must have a negative blood pregnancy test at Screening, and if randomized to vaccination a negative blood or urine pregnancy test within one (1) day before each dose of Intuvax, or Male agreeing to use condoms during the study participation or male having a female partner who is using a highly efficient method of contraception as described above during the partner's study participation.

Exclusion Criteria:

1. Performance status > ECOG 2
2. Known major reaction/adverse event in connection with previously made vaccination (e.g. asthma, anaphylaxia or other serious reaction)
3. Known major reaction/adverse event in connection with previous transfusions of blood products
4. Active autoimmune disease requiring treatment with systemic immunosuppressive agents, e.g. inflammatory bowel disease, multiple sclerosis, sarcoidosis, psoriasis, autoimmune hemolytic anemia, rheumatoid arthritis, SLE, vasculitis, Sjögren's syndrome, scleroderma, autoimmune hepatitis, and other rheumatological diseases.
5. Tested positive for HIV
6. Active virus disease (HBV and HCV).
7. Ongoing infection that requires treatment with parenteral antibiotics or antiviral medication
8. Corticosteroid treatment per os exceeding 10mg/day within 7 days prior to the first injection of Intuvax. Inhaled, intranasal and local steroids accepted.
9. Inadequate laboratory parameters, i.e.:

   * B-Leukocyte count < 3.0 x109/L
   * B-Platelet count < 75 x109/L
   * B-Hemoglobin < 100 g/L
   * P-Prothrombincomplex (PK) >1.4
   * P-APT time outside normal limit
10. Previous organ transplantation
11. Pregnant or lactating women
12. Life expectancy less than 3 months.
13. Investigational treatment (within 28 days) prior to the first injection of Intuvax
14. Known blood dyscrasia (bleeding complication)
15. Prior history of invasive cancer within 5 years before screening, except for adequately treated in situ carcinomas or non melanoma skin cancer
16. History of alcohol or substance abuse
17. patient will not be available for follow up assessments
18. Any other reason that, in the opinion of the investigator, contraindicates that the patient participates in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Changes in vital signs (heart rate, blood pressure, body temperature) | Up to 12 months after vaccination 1
Changes in lab parameters (hematology and biochemistry) during the study versus baseline | Up to 12 months after vaccination 1
Adverse events according to CTCAE v 4.03 | Up to 12 months after vaccination 1

SECONDARY OUTCOMES:
Tumor response by determining changes (PD, SD, PR, CR) in tumor diameter according to mRECIST | Every 3 months up to 12 months after vaccination 1
  Criteria based on the diameter of the contrast-enhanced portions of the tumor
Tumor response by determining changes (PD, SD, PR, CR) in tumor diameter according to RECIST 1.1. | Every 3 months up to 12 months after vaccination 1
  Criteria based on the maximal tumor diameter
Tumor response by determining changes (PD, SD, PR, CR) in tumor diameter according to Choi criteria | Every 3 months up to 12 months after vaccination 1
  Criteria based on unidimensional tumor size and tumor density on contrast-enhanced CT images.
Progression free survival according to mRECIST | Up to 12 months after vaccination 1
  Criteria based on the diameter of the contrast-enhanced portions of the tumor
Progression free survival according to RECIST 1.1 | Up to 12 months after vaccination 1
  Criteria based on the maximal tumor diameter
Progression free survival according to Choi criteria | Up to 12 months after vaccination 1
  Criteria based on unidimensional tumor size and tumor density on contrast-enhanced CT images.
Changes in WHO-ECOG score | Up to 12 months after vaccination 1
Levels of autoimmunization parameters | Up to 3 months after vaccination 1
  Screening of autoantibodies against nuclear antigens (ANA), including the nuclear antigens SSA, SSB, Sm, RNP, Scl-70, Centromeres and Jo-1
Levels of alloimmunization parameters | Up to 3 months after vaccination 1
  Screening of alloantibodies against HLA-A, B, C (MHC-class I) and HLA-DR (MHC-class II) antigens

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mendus
Locations (1):
- Department of Breast and Endocrine Surgery, Section of Endocrine and Sarcoma Surgery, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No